CLINICAL TRIAL: NCT05840510
Title: A Phase 1/2 Trial of Adagrasib in Combination With Nab-Sirolimus in Patients With Advanced Solid Tumors and Non-Small Cell Lung Cancer With a KRAS G12C Mutation
Brief Title: Adagrasib in Combination With Nab-Sirolimus in Patients With Advanced Solid Tumors and Non-Small Cell Lung Cancer With a KRAS G12C Mutation (KRYSTAL -19)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Mirati Therapeutics Inc. (Industry)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0011; CA239-0011 (Other: Bristol-Myers Squibb Protocol ID); 849-019 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor, Adult; NSCLC; Advanced Cancer; Metastatic Cancer; Malignant Neoplastic Disease
Keywords: KRAS; NSCLC; Adagrasib; KRAS G12C; mTOR; nab-sirolimus; Fyarro; ABI-009
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Clinical Efficacy (Experimental): Dose escalation of adagrasib and nab-Sirolimus to determine maximum tolerated dose in combination and evaluate the clinical efficacy of adagrasib in combination with nab-sirolimus in patients with solid tumors (Phase 1) and NSCLC (Phase 2) harboring a KRAS G12C mutation
  Interventions: Drug: Adagrasib; Drug: nab-Sirolimus

INTERVENTIONS:
Drug: Adagrasib — KRAS G12C inhibitor
  Other Names: MRTX849; Krazati
Drug: nab-Sirolimus — mTOR inhibitor
  Other Names: ABI -009; Fyarro

SUMMARY:
This study will evaluate the safety, MTD and/or RP2D, PK, and clinical activity of the combination of adagrasib with nab-sirolimus in patients with advanced solid tumors/NSCLC with a KRAS G12C mutation.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability and clinical activity of adagrasib in combination with nab-sirolimus in patients with advanced solid tumors harboring a KRAS G12C mutation.

The Phase 1 portion will enroll advanced solid tumors to establish the maximum tolerated dose (MTD) and/or to identify recommended Phase 2 combinatorial doses. The Phase 2 portion will enroll patients with NSCLC to further evaluate the safety/tolerability and clinical activity.

Adagrasib is an orally available small molecule inhibitor of KRAS G12C. nab-Sirolimus is a nanoparticle albumin-bound (nab) form of sirolimus, and sirolimus is an inhibitor of mechanistic target of rapamycin kinase (mTOR, previously known as mammalian target of rapamycin).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of solid tumor malignancy (Phase 1) or NSCLC (Phase 2) with KRAS G12C mutation
* Unresectable or metastatic disease
* No available treatment with curative intent
* Adequate organ function
* Measurable disease per RECIST 1.1.

Exclusion Criteria:

* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow
* History of interstitial lung disease or radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease or pneumonitis
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability in the study population. | 30 months
  Safety characterized by the following, as noted from first dose of study treatment to 28 days after last dose of study treatment:
  1. Type, incidence, severity, timing, seriousness and relationship to study treatment of Adverse Events
  2. Laboratory abnormalities, as measured by changes in lab results such as hematologic or chemistry parameters while on study treatment
  3. Number of patients modifying or discontinuing study treatment due to an AE
Phase 1: Maximum tolerated dose (MTD) and Recommended Phase 2 Dose (RP2D) | 30 months
  Evaluate safety and assess number of patients with dose-limiting toxicity to determine the MTD/RP2D.
Phase 2: Objective Response Rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) (Phase 2) | 30 months
  ORR evaluation of subjects treated with adagrasib in combination with nab-sirolimus in patients with NSCLC with KRAS G12C mutation (Study Population) will be completed. Objective response is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from first dose of study treatment until last dose of study treatment.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 7 days
  AUC - nab-sirolimus and adagrasib
Time to achieve maximal plasma concentration | Up to 1 days
  Tmax - nab-sirolimus and adagrasib
Maximum observed plasma concentration | Up to 1 days
  Cmax - nab-sirolimus and adagrasib
Terminal elimination half-life | Up to 7 days
  t1/2 - nab-sirolimus
Phase 1 and 2: Evaluate efficacy endpoints characterized by overall survival, progression-free survival, and duration of response in the study population. | 30 months
  1. Overall survival is defined as time from date of randomization to date of death due to any cause.
  2. Progression-free survival is defined as the time from randomization to the date of Progressive Disease (PD) or death due to any cause,whichever occurs first.
  3. Duration of response defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either PD or death due to any cause, whichever occurs first.
Phase 1: Objective Response Rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) | 30 months
  ORR evaluation of subjects treated with adagrasib in combination with nab-sirolimus in patients with advanced solid tumors and NSCLC with KRAS G12C mutation (Study Population) will be completed. Objective response is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from first dose of study treatment until last dose of study treatment.
Phase 2: Safety and tolerability in the study population. | 30 months
  Safety characterized by the following, as noted from first dose of study treatment to 28 days after last dose of study treatment:
  1. Type, incidence, severity, timing, seriousness and relationship to study treatment of Adverse Events
  2. Laboratory abnormalities, as measured by changes in lab results such as hematologic or chemistry parameters while on study treatment
  3. Number of patients modifying or discontinuing study treatment due to an AE,

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 019-104, Cleveland, Ohio
  - Local Institution - 019-101, Nashville, Tennessee
  - Local Institution - 019-102, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com